CLINICAL TRIAL: NCT05338723
Title: Possible Protective Effect of Rosuvastatin in Chemotherapy-induced Cardiotoxicity in HER2 Positive Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Khlood Mohamed Kettana, demonstrator at clinical pharmacy department,faculty of pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: rosuva2020
Record Dates: First submitted 2022-04-04; First posted 2022-04-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chemotherapy-induced Cardiotoxicity; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control-group (No Intervention): This group will include 25 patients who will receive doxorubicin for 4 cycles (3 months) followed by trastuzumab adjuvant therapy.
- rosuvastatin-group (Active Comparator): This group will include 25 patients who will receive doxorubicin for 4 cycles (3 months) followed by trastuzumab adjuvant therapy in addition to 20 mg of oral rosuvastatin 24 hours prior to the first cycle of chemotherapy and once daily for the rest of the follow-up period (6 months).
  Interventions: Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Rosuvastatin 20mg — 20 mg of oral rosuvastatin 24 hours prior to the first cycle of chemotherapy and once daily for the rest of the follow-up period (6 months).
  Arms: rosuvastatin-group

SUMMARY:
This study aims to investigate the possible role of rosuvastatin in protection against cardiotoxicity in HER2 positive breast cancer patients receiving doxorubicin sequential with trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-75 years old.
* Gender: female
* Newly diagnosed HER2 positive breast cancer patients who are scheduled to receive doxorubicin followed by trastuzumab adjuvant therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
* Preserved LV systolic function in which the left ventricular ejection fraction (LVEF)≥50%.
* Patients with normal renal and hematological functions.
* Alanine amino transferase (ALT ≤ 3 times ULN).

Exclusion Criteria:

* Pregnant or lactating females.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) > 2
* Patients with impaired LV systolic function in which the left ventricular ejection fraction (LVEF)<50%.
* Patients with significant valvular heart disease, documented coronary artery disease, history of congestive heart failure or cardiomyopathy.
* Alanine amino transferase (ALT > 3 times ULN).
* Patients already taking statins or other lipid lowering therapy.
* Patients with a known hypersensitivity to any of the used drugs.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only female patients are included in the study
Enrollment: 50 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
change in left ventricular ejection fraction(LVEF) detected by electrocardiography transthoracic echocardiography | 6 months
  Patients will undergo transthoracic echocardiography 24 hours prior to the initiation of chemotherapy, after 3 months and after 6 months to detect change in LVEF

SECONDARY OUTCOMES:
change of serum level of High sensitivity troponin I (hs-TnI). | 6 months
  Blood samples will be collected at baseline, after 3 months and after 6 months to evaluate High sensitivity troponin I (hs-TnI).
change of serum level of Myeloperoxidase (MPO). | 6 months
  Blood samples will be collected at baseline, after 3 months and after 6 months to evaluate Myeloperoxidase (MPO).
change of serum level of Interleukin-6 (IL-6). > Liver function test (ALT). | 6 months
  Blood samples will be collected at baseline, after 3 months and after 6 months to evaluate Interleukin-6 (IL-6).
change of serum level of Liver function test (ALT). | 6 months
  Blood samples will be collected at baseline, after 3 months and after 6 months to evaluate Liver function test (ALT).

CONTACTS AND LOCATIONS:
Overall Officials: khlood m. kettana, Principal Investigator — Tanta University
Locations (1):
- The Department of Clinical Oncology, Tanta University Hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No